CLINICAL TRIAL: NCT01796964
Title: A Prospective, Randomized, Double-Masked, Multicenter, Two Arm Study Comparing the Efficacy and Safety of ESBA1008 Versus EYLEA® in Subjects With Exudative Age-Related Macular Degeneration
Brief Title: Efficacy and Safety Study of ESBA1008 Versus EYLEA®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-12-006
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Wet; Exudative; AMD; Intravitreal injection; Retina
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESBA1008 (Experimental): ESBA1008 solution, 7 intravitreal (IVT) injections, as specified in protocol
  Interventions: Drug: ESBA1008 solution
- EYLEA (Active Comparator): Aflibercept, 8 intravitreal (IVT) injections, as specified in protocol
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: ESBA1008 solution — For intravitreal (IVT) injection
  Arms: ESBA1008
Drug: Aflibercept — For intravitreal (IVT) injection
  Other Names: EYLEA®
  Arms: EYLEA

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ESBA1008 versus EYLEA® in the treatment of exudative age-related macular degeneration.

DETAILED DESCRIPTION:
This study consisted of 16 visits (Screening, Baseline [Day 0], and 14 post-baseline assessment visits) that occurred at 4-week intervals through Week 56. Enrolled subjects were randomized 1:1 to receive ESBA1008 or EYLEA. All subjects received active intravitreal (IVT) injections at baseline with 2 additional loading doses of the assigned investigational product at 4-week intervals (ie, at Weeks 4 and 8) and then received further injections at 8-weeks intervals at Weeks 16, 24, and 32. Subjects in the ESBA1008 group also received an injection at Week 44, while subjects in the EYLEA group also received injections at Weeks 40 and 48. To maintain the study masking, subjects in the ESBA1008 group received sham injections at Weeks 40 and 48 (when the subjects in the EYLEA group received active injections), while subjects in the EYLEA group received a sham injection at Week 44 (when the subjects in the ESBA1008 group received an active injection). All subjects were followed up to Week 56. Week 40 visit was the end of assessment period for the 8-week treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent; be able to make the required study visits and follow instructions.
* Diagnosis of wet age-related macular degeneration, as specified in protocol.
* Best-corrected visual acuity (BCVA) as specified in protocol
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Either eye: Any active ocular or periocular infection or active intraocular inflammation.
* Study eye: Any approved or investigational treatment for exudative AMD other than vitamin supplements.
* Study eye: Any current or history of macular or retinal disease other than exudative AMD.
* Study eye: Any concurrent intraocular condition that, in the opinion of the Investigator, could require medical or surgical intervention during the course of the study to prevent or treat vision loss, or that limits the potential to gain visual acuity with the investigational product.
* Study eye: Uncontrolled glaucoma.
* Study eye: Any ocular disease that, in the opinion of the Investigator, could compromise the visual acuity.
* Study eye: History of eye surgery, as specified in protocol.
* Study eye: Use of corticosteroids, as specified in protocol.
* Any medical condition that, in the opinion of the Investigator, would preclude scheduled study visits, completion of the study or safe administration of investigational product.
* Any screening laboratory result that, in the opinion of the Investigator, would make the patient unsuitable for study participation.
* History of hypersensitivity to any component used in the study, as assessed by the Investigator.
* Women of childbearing potential: Lactating, pregnant, plan to become pregnant, or not using adequate birth control, as specified in protocol.
* Participation in an investigational drug or device study within time period specified in protocol.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Pharma, Study Director — Alcon Research

REFERENCES:
- [Derived] Dugel PU, Jaffe GJ, Sallstig P, Warburton J, Weichselberger A, Wieland M, Singerman L. Brolucizumab Versus Aflibercept in Participants with Neovascular Age-Related Macular Degeneration: A Randomized Trial. Ophthalmology. 2017 Sep;124(9):1296-1304. doi: 10.1016/j.ophtha.2017.03.057. Epub 2017 May 24. PMID 28551167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 41 investigational centers located in the US.
Pre-assignment Details: Of the 173 enrolled, 83 subjects were exited as screen failures prior to randomization. One randomized subject did not receive treatment. Another subject randomized to ESBA 1008 received EYLEA treatment. This reporting group includes all randomized and treated subjects, as treated (ESBA1008: 44 subjects and EYLEA: 45 subjects).
Period: Overall Study
Arm/Group | ESBA1008 | EYLEA
Started | 44 | 45
Completed | 41 | 42
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized, received at least 1 treatment, had a baseline value, and had at least 1 postbaseline measurement of the primary efficacy variable, BCVA. Subjects were analyzed according to the actual treatment received with last observation carried forward (LOCF) imputation of missing values.
Groups:
- Total: Total of all reporting groups
Arm/Group | ESBA1008 | EYLEA | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.8 (9.7) | 77.3 (9.1) | 78.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Best-Corrected Visual Acuity (BCVA) Change From Baseline (No. of Letters) to Week 12
Description: This outcome measure was used to compare the ESBA1008 and EYLEA groups in regards to fluctuations in treatment effect during the maintenance phase with 8-week treatment cycles (ie, to evaluate treatment effect stability during the maintenance phase). BCVA (with spectacles or other visual corrective devices) using Early Treatment Diabetic Retinopathy Study (ETDRS) testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 12
Population: This analysis population includes all subjects who were randomized, received at least 1 treatment, had a baseline value, and had at least 1 postbaseline measurement of the primary efficacy variable, BCVA. Subjects were analyzed according to the actual treatment received with LOCF imputation of missing values.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Baseline (Day 0) | 54.1 (13.9) | 55.6 (12.3)
  Change from baseline | 5.8 (12.7) | 6.9 (9.3)
Statistical Analysis 1: Comparison: ESBA1008 vs EYLEA; An analysis of variance (ANOVA) model with treatment and baseline BCVA categories (< 55 and ≥ 55 letters) as class variables was used to estimate the treatment group differences (ESBA1008 - EYLEA) in the primary efficacy endpoint, BCVA Change from baseline to Week 12; Test type: Non-Inferiority or Equivalence — Non-inferiority at week 12 is concluded at one-sided alpha level of 0.10 if the lower limit of the corresponding two-sided 80% confidence interval for the treatment difference (ESBA 1008 - EYLEA) is greater than -5 letters; Treatment difference (ESBA - Eylea) = -1.13, 80% CI 2-sided [-4.19 to 1.93] — Treatment differences were based on least squares estimates

2. Secondary Outcome: BCVA Change From Baseline (No. of Letters) to Week 16
Description: BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Baseline (Day 0) | 54.1 (13.9) | 55.6 (12.3)
  Change from baseline | 6.0 (13.3) | 6.6 (9.2)
Statistical Analysis 1: Comparison: ESBA1008 vs EYLEA; An analysis of variance (ANOVA) model with treatment and baseline BCVA categories (< 55 and ≥ 55 letters) as class variables was used to estimate the treatment group differences (ESBA1008 - EYLEA) in the primary efficacy endpoint, BCVA Change from baseline to Week 16; Test type: Non-Inferiority or Equivalence — Non-inferiority at week 16 is concluded at one-sided alpha level of 0.10 if the lower limit of the corresponding two-sided 80% confidence interval for the treatment difference (ESBA 1008 - EYLEA) is greater than -5 letters; Treatment difference (ESBA - Eylea) = -0.58, 80% CI 2-sided [-3.72 to 2.56] — Treatment differences were based on least squares estimates

3. Secondary Outcome: BCVA Change From Baseline (No. of Letters) by Visit
Description: as for outcome 2
Time Frame: Baseline (Day 0), Week 4, Week 8, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Baseline (Day 0) | 54.1 (13.9) | 55.6 (12.3)
  Change from baseline at Week 4 | 4.8 (9.1) | 4.3 (7.4)
  Change from baseline at Week 8 | 6.0 (11.6) | 6.5 (8.5)
  Change from baseline at Week 20 | 7.5 (14.5) | 7.3 (9.4)
  Change from baseline at Week 24 | 7.1 (13.0) | 8.2 (11.2)
  Change from baseline at Week 28 | 8.3 (12.2) | 6.6 (12.4)
  Change from baseline at Week 32 | 6.7 (13.7) | 6.5 (12.7)
  Change from baseline at Week 36 | 6.2 (16.2) | 6.4 (13.1)
  Change from baseline at Week 40 | 6.3 (14.9) | 5.7 (13.6)
  Change from baseline at Week 44 | 7.0 (15.6) | 6.5 (12.0)
  Change from baseline at Week 48 | 6.2 (16.5) | 6.8 (13.4)
  Change from baseline at Week 52 | 6.0 (16.4) | 7.2 (13.2)
  Change from baseline at Week 56 | 4.9 (17.9) | 7.3 (13.4)

4. Secondary Outcome: Average BCVA Change From Baseline (No. of Letters) Over the Periods of Week 4 to Week 16, Week 4 to Week 24, Week 4 to Week 40, and Week 4 to Week 56
Description: The purpose of this outcome measure was to assess the integrated effect of the treatment for different study periods and to provide more robust estimate of the absolute treatment effects. BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. These changes were computed as the average of the changes from baseline to each monthly study visit corresponding to each period. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Baseline (Day 0) | 54.1 (13.9) | 55.6 (12.3)
  Avg Change from baseline over period of Weeks 4-16 | 5.7 (11.0) | 6.1 (8.0)
  Avg Change from baseline over period of Weeks 4-24 | 6.2 (11.7) | 6.6 (8.4)
  Avg Change from baseline over period of Weeks 4-40 | 6.5 (12.3) | 6.5 (9.2)
  Avg Change from baseline over period of Weeks 4-56 | 6.4 (13.3) | 6.6 (10.0)

5. Secondary Outcome: Average BCVA Change From Week 12 (No. of Letters) Over the Periods of Week 16 to Week 24, Week 16 Week 40, and Week 16 to Week 56
Description: The purpose of this outcome measure was to assess the average maintenance level of BCVA following the 3 loading treatments (ie, after Week 12). BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. These changes were computed as the average of the changes from Week 12 to each monthly study visit corresponding to each period. One eye (study eye) contributed to the analysis.
Time Frame: Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Week 12 | 59.8 (18.5) | 62.4 (16.1)
  Avg Change from Week 12 over period Weeks 16-24 | 1.1 (5.4) | 0.5 (4.7)
  Avg Change from Week 12 over period Weeks 16-40 | 1.1 (6.3) | -0.1 (7.3)
  Avg Change from Week 12 over period Weeks 16-56 | 0.8 (7.0) | -0.0 (8.1)

6. Secondary Outcome: One-Month BCVA Changes (No. of Letters) Following No Treatment for 1-Month
Description: The purpose of this outcome measure was to assess the stability of BCVA during the second month of 8-week/12-week treatment cycles and specifically to identify potential under treatment. BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Change from Week 12 to Week 16 | 0.3 (5.7) | -0.2 (5.1)
  Change from Week 20 to Week 24 | -0.4 (4.8) | 0.9 (5.5)
  Change from Week 28 to Week 32 | -1.7 (4.6) | -0.1 (3.6)
  Change from Week 36 to Week 40 | 0.1 (7.3) | -0.7 (4.0)
  Change from Week 44 to Week 48 | NA (NA) — Subjects in the ESBA1008 group received active IVT injections at Day 0 and at Weeks 4, 8, 16, 24, 32, and 44. | 0.2 (4.2)
  Change from Week 48 to Week 52 | -0.1 (4.3) | NA (NA) — Subjects in the EYLEA group received IVT injections at Day 0, Weeks 4, 8, 16, 24, 32, 40, and 48.
  Change from Week 52 to Week 56 | NA (NA) — Subjects in the ESBA1008 group received active IVT injections at Day 0 and at Weeks 4, 8, 16, 24, 32, and 44. | 0.0 (4.2)

7. Secondary Outcome: One-Month BCVA Changes (No. of Letters) Following Treatment by Visit
Description: The purpose of this outcome measure was to assess the potential treatment needs present at these treatment visits. BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
letters
  Change from Week 16 to Week 20 | 1.5 (5.7) | 0.6 (5.1)
  Change from Week 24 to Week 28 | 1.2 (5.6) | -1.6 (7.7)
  Change from Week 32 at Week 36 | -0.5 (7.9) | -0.2 (5.1)
  Change from Week 40 to Week 44 | NA (NA) — Subjects in the ESBA1008 group received active IVT injections at Day 0 and at Weeks 4, 8, 16, 24, 32, and 44. | 0.8 (5.2)
  Change from Week 44 to Week 48 | -0.8 (4.2) | NA (NA) — Subjects in the EYLEA group received IVT injections at Day 0, Weeks 4, 8, 16, 24, 32, 40, and 48.
  Change from Week 48 to Week 52 | NA (NA) — Subjects in the ESBA1008 group received active IVT injections at Day 0 and at Weeks 4, 8, 16, 24, 32, and 44. | 0.5 (3.6)

8. Secondary Outcome: Two-Months BCVA Changes (No. of Letters) Following No Treatment for 1 Month in ESBA Treatment Group
Description: BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. This outcome measure was pre-specified for ESBA1008 arm only. One eye (study eye) contributed to the analysis.
Time Frame: Week 36, Week 44, Week 48, Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | ESBA1008
Number analyzed (Participants) | 44
letters
  Change from Week 36 to Week 44 | 0.8 (7.1)
  Change from Week 48 to Week 56 | -1.3 (5.0)

9. Secondary Outcome: Central Subfield Thickness (CSFT) Change From Baseline by Visit
Description: CSFT (average thickness in the central subfield centered at the fovea) as measured using Spectral-Domain Optical Coherence Tomography (SD-OCT). Reduction in CSFT measurement from baseline indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ESBA1008 | EYLEA
Number analyzed (Participants) | 44 | 45
microns
  Baseline (Day 0) | 490.1 (149.2) | 495.7 (144.6)
  Change from baseline at Week 4 | -184.7 (118.9) | -153.0 (95.1)
  Change from baseline at Week 8 | -198.5 (117.6) | -176.1 (106.5)
  Change from baseline at Week 12 | -199.5 (126.7) | -186.2 (113.6)
  Change from baseline at Week 16 | -188.4 (121.0) | -163.2 (116.4)
  Change from baseline at Week 20 | -207.0 (123.2) | -184.8 (118.5)
  Change from baseline at Week 24 | -194.0 (127.9) | -164.0 (121.8)
  Change from baseline at Week 28 | -210.0 (125.0) | -185.9 (117.9)
  Change from baseline at Week 32 | -205.8 (124.3) | -166.4 (123.2)
  Change from baseline at Week 36 | -213.0 (132.4) | -185.3 (117.7)
  Change from baseline at Week 40 | -200.6 (143.6) | -175.2 (124.1)
  Change from baseline at Week 44 | -196.1 (120.2) | -184.6 (121.7)
  Change from baseline at Week 48 | -213.0 (129.7) | -175.7 (124.3)
  Change from baseline at Week 52 | -210.5 (130.6) | -198.8 (123.4)
  Change from baseline at Week 56 | -196.8 (135.4) | -180.4 (121.6)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 56 weeks). AEs were reported as pre-treatment and treatment-emergent. Ocular AEs are presented for both study eye and non-study eye combined.
Description: An AE was defined as any untoward medical occurrence in a subject administered a study treatment regardless of causal relationship. AEs were obtained as solicited comments from the study subjects and as observations by the study Investigator.
Groups:
- Pre-treatment: All subjects who consented to participate in the study
- ESBA 1008: All subjects who were randomized and received at least 1 IVT injection of ESBA1008 solution
- EYLEA: All subjects who were randomized and received at least 1 IVT injection of Aflibercept
Arm/Group | Pre-treatment | ESBA 1008 | EYLEA
Serious Adverse Events (participants affected / at risk) | 0/173 | 11/44 | 9/45
Other Adverse Events (participants affected / at risk) | 0/173 | 22/44 | 25/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=173) | ESBA 1008 (N=44) | EYLEA (N=45)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=173) | ESBA 1008 (N=44) | EYLEA (N=45)
Age-related macular degeneration (Eye disorders) | 0 | 5 | 2 — ESBA: Two subjects experienced AEs in the non-study eye; EYLEA: One subject experienced an AE in the non-study eye
Cataract (Eye disorders) | 0 | 1 | 3
Conjunctival haemorrhage (Eye disorders) | 0 | 5 | 7
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 3
Macular fibrosis (Eye disorders) | 0 | 3 | 1
Punctate keratitis (Eye disorders) | 0 | 2 | 3 — ESBA: One subject experienced an AE in the non-study eye
Retinal haemorrhage (Eye disorders) | 0 | 2 | 3
Vision blurred (Eye disorders) | 0 | 2 | 3 — ESBA: One subject experienced an AE in the non-study eye
Visual acuity reduced (Eye disorders) | 0 | 5 | 4 — ESBA: One subject experienced an AE in the non-study eye
Vitreous detachment (Eye disorders) | 0 | 3 | 4 — EYLEA: One subject experienced an AE in the non-study eye
Vitreous floaters (Eye disorders) | 0 | 5 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.